CLINICAL TRIAL: NCT05424770
Title: The Effect of Crossword Used as an Active Learning Tool in Nursing Education on Learning Achievement: A Randomized Controlled Study
Brief Title: The Effect of the Crossword Used in Nursing Education on Learning Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Sevgi Deniz Dogan, lecturer Dr., Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 5312256942
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Pain; Nursing; Crossword
MeSH Terms: conditions — Pain | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental): During the 3 weeks in which the subjects related to pain control are explained, the standard lecture (explanation with ppt presentation) will be made as in the normal course of the course. Afterwards, puzzle activities prepared by the researcher will be implemented and students will be actively involved in the process.
  Interventions: Other: Education with crossword
- control group (No Intervention): During the 3 weeks in which the subjects related to pain control are explained, the standard lecture (explanation with ppt presentation) will be made as in the normal course of the course.

INTERVENTIONS:
Other: Education with crossword — Afterwards, crossword activities prepared by the researcher will be implemented and students will be actively involved in the process. The researcher will also include a collaborative learning environment where students can exchange information with each other. After the completion of each puzzle, the researcher will make the necessary checks and corrections.
  Arms: experiment group

SUMMARY:
The research was planned as a randomized controlled study to evaluate the effect of crossword, which are an active learning tool, on the success of learning information about pain control in nursing education. Research data is planned to be collected in Hatay Mustafa Kemal University Faculty of Health Sciences. The universe of the research will be the students who take the 3-credit pain control course in the aforementioned faculty in the fall semester. The sample of the research will consist of 72 students who meet the inclusion criteria and agree to participate in the research verbally and in writing. The data of the research will be collected by using the Personal information form prepared in line with the literature, and Success Tests (3 tests) prepared separately for each stage. SPSS program will be used in the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* To be registered in the pain course,
* Taking the pain course for the first time,
* Absence of any psychiatric disorder that will reduce the ability to comprehend and understand,
* Agreeing to participate in the research.

Exclusion Criteria:

-Willingness to leave the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The effect of crossword on learning achievement in nursing education | Three months
  Evaluation will be made with a multiple-choice (5-choice) achievement test, which will be prepared by the researchers within the scope of the application. This test will consist of 20 items. After the test is prepared, item analysis will be made and it will be presented to the expert opinion. In the test, each correct answer will be scored as 1 and each incorrect answer as 0. The higher the score, the higher the success will be interpreted.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University Institute of Health Sciences, Hatay, Turkey (Türkiye)

REFERENCES:
- [Derived] Kose Tosunoz I, Deniz Dogan S. The effect of crossword puzzles on nursing students' learning of concepts related to pain management course: A randomized controlled trial. Nurse Educ Pract. 2023 Aug;71:103740. doi: 10.1016/j.nepr.2023.103740. Epub 2023 Aug 3. PMID 37544239